CLINICAL TRIAL: NCT04366258
Title: Transcranial Near Infrared Radiation and Cerebral Blood Flow in Depression
Acronym: TRIADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-00217; 1R61MH122647-01 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-04-28 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder
Keywords: MDD, neuromodulation, transcranial photobiomodulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with MDD (Experimental): Participants will undergo 4 Transcranial Photobiomodulation (t-PBM) treatment visits and receive 1 irradiance dose per visit. The order of dose administration is randomized so patients receive each irradiance dose (50 mW/cm2; 300 mW/cm2; 770 mW/cm2), as well as a sham dose (0 mW/cm2), once over the 4 treatment visits.
  Interventions: Device: Transcranial Photobiomodulator; Device: Sham

INTERVENTIONS:
Device: Transcranial Photobiomodulator — Delivers laser-generated Near-Infrared Radiation (NIR) to forehead at 3 doses of irradiance - High (770 mW/cm2), Middle (300 mW/cm2), and Low (50 mW/cm2).
  Other Names: LightForce® EXPi Deep Tissue Laser TherapyTM System, Transcranial PhotoBioModulation-1000 (tPBM-2.0)
Device: Sham — Transcranial Photobiomodulator delivers sham irradiance dose of 0 mW/cm2.

SUMMARY:
This study will compare the effect of three transcranial photobiomodulation (t-PBM) doses (high, middle, and low irradiance) to sham t-PBM on PFC CBF as assessed with fMRI (BOLD) in this multi-center, phase I, double-blinded, dose-ranging, controlled, crossover study of 30 subjects with MDD. All eligible participants will undergo four sessions of t-PBM during fMRI so that they experience irradiances of 50, 300 and 700 mW/cm2 as well as sham. The order of dose administration will be randomized and t-PBM will be administered with the LightForce® EXPi Deep Tissue Laser TherapyTM System, Transcranial PhotoBioModulation-1000 (tPBM-2.0).

DETAILED DESCRIPTION:
The purpose of this research study is to determine if application of near infrared energy to the forehead can change blood flow in the brains of people with depression. Near infrared energy is like light but is not visible to the human eye. This research study will compare near infrared exposure with a placebo or sham procedure. The sham procedure will look and feel just like the near infrared procedure but won't include near infrared exposure.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to give written informed consent and follow study procedures
* Participants must have major depressive disorder; all the following conditions need to be met to ensure presence of significant depression symptoms:

  1. Meeting diagnostic criteria for Major Depressive Disorder (MDD) in the past two weeks, at the DSM-5 Mini-International Neuropsychiatric Interview (MINI)
  2. Inventory for Depressive Symptomatology Clinician-rated (IDS-C) total score ≥23 at screening
  3. Depression symptoms are the primary target of treatment or treatment-seeking.
* Women of child-bearing potential must agree to use adequate contraception
* Participants taking medications or psychotherapy approved for the treatment of major depressive disorder will need to be stable for at least 8 weeks prior to screen

Exclusion Criteria:

* Unwilling or unable to comply with study requirements
* Participants who are judged to be at serious and imminent suicidal (C-SSRS≥4) or homicide risk, or currently in crisis such that inpatient hospitalization or other crisis management should take priority
* History of any or psychotic or bipolar disorder
* Alcohol or substance use disorder, post-traumatic stress disorder, obsessive-compulsive disorder and eating disorders within the preceding 12 months
* History of dementia, traumatic brain injury (TBI), or neurological disorders affecting the brain, including any history of stroke or seizure disorders requiring treatment in the last 5 years (even if controlled with medications)
* Cognitive impairment significant as determined by the Montreal Cognitive Assessment (MOCA) <22
* History of antisocial personality disorder, or any clinically significant personality trait that would, in the investigator's judgment, preclude safe study participation or impair ability to remain adherent with the treatment protocol.
* History of significant treatment non-adherence or situations where the subjects are unlikely to adhere to treatment, in the opinion of the investigator
* Pregnant (as confirmed by pregnancy test at screen) or nursing.
* Currently undergoing device-based treatment for depression or taking medications for depression other than SSRIs or SNRIs.
* Treatment resistance with failure to respond to more than two adequate treatments with FDA-approved antidepressant medications during current episode of major depressive disorder.
* History of ECT in the last 12 months; lifetime history of VNS; lifetime treatment resistance to any FDA-approved device-based treatment for major depressive disorder; device-based interventions for depression will need to be discontinued at least 8 weeks prior to screen.
* Serious, unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, hematologic disease; defined as any medical illness which is not well-controlled with standard-of-care medications
* Clinically significant abnormal findings of laboratory parameters including urine toxicology screen for drugs of abuse or at physical examination
* Clinical or laboratory evidence of uncontrolled hypothyroidism; if maintained on thyroid medication must be euthyroid for at least 1 month before screening.
* Past intolerance or hypersensivity to t-PBM.
* Significant skin conditions on the subject's scalp that are found in the area of the procedure sites.
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.
* Any type of implants in the head, whose functioning might be affected by t-PBM.
* Failure to meet standard MRI safety requirements as determined by the MRI Safety Checklist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - New York University, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and upon reasonable request. Requests should be directed to Dr. Kate Collins, PhD (email: Kate.Collins@nki.rfmh.org). To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The cross-over study enrolled 55 participants. The 31 participants who met study criteria were assigned to receive 4 irradiance dose levels of t-PBM in random order across 4 t-PBM sessions (1 dose per session, doses assigned in random order: t-PBM at High Irradiance, t-PBM at Middle Irradiance, t-PBM at Low Irradiance, and Sham).
Groups:
- Patients With MDD: Participants underwent 4 Transcranial Photobiomodulation (t-PBM) treatment visits and received 1 irradiance dose per visit. The order of dose administration is randomized so patients receive each irradiance dose (50 mW/cm2; 300 mW/cm2; 770 mW/cm2), as well as a sham dose (0 mW/cm2), once over the 4 treatment visits.
Period: Baseline Assessments
Arm/Group | Patients With MDD
Started | 55
Completed | 31
Not Completed | 24
Not completed — Screen Failure | 21
Not completed — Early Termination | 3
Period: Randomized Cross-Over
Arm/Group | Patients With MDD
Started | 31
Received t-PBM at High Irradiance | 27
Received t-PBM at Medium Irradiance | 29
Received t-PBM at Low Irradiance | 29
Received t-PBM at Sham Irradiance | 29
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristic information was collected from 30 of the 31 participants who completed the baseline period and were assigned to treatment.
Groups:
- Overall Study Population: All participants from whom baseline characteristics were collected.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.08 (15.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Prefrontal Cortex (PFC) Cerebral Blood Flow (CBF) During High-Irradiance t-PBM
Description: CBF is measured as Blood Oxygen Level Dependent (BOLD) signal on functional magnetic resonance imaging (fMRI). BOLD signal reflects changes in regional CBF that delineate regional activity. A positive BOLD signal marks an increase in regional blood flow, while a negative BOLD signal marks a decrease in regional blood flow. A positive percent change indicates that blood flow increased in the region of interest between scans, a negative percent change indicates blood flow decreased between scans.
  Approximately 60 minutes of fMRI data are recorded in the left and right dorsolateral prefrontal cortical regions of interest at each transcranial photobiomodulation (t-PBM) treatment visit, including: approximately 20 minutes prior to t-PBM administration, approximately 20 minutes coinciding with t-PBM administration, and approximately 20 minutes following t-PBM administration.
Time Frame: 20 Minutes Pre-Intervention, 20 Minutes Post-Intervention (Total duration: 60 min); Up to Week 7
Measure: Mean (Standard Deviation); unit: Percent change in raw frontal BOLD
Groups:
- t-PBM at High Irradiance: At 1 of the 4 t-PBM sessions, participants were administered t-PBM at high irradiance (at least 700 mW/cm2).
Arm/Group | t-PBM at High Irradiance
Number analyzed (Participants) | 27
Percent change in raw frontal BOLD | 1.12 (25.07)

2. Primary Outcome: Percentage Change in Prefrontal Cortex (PFC) Cerebral Blood Flow (CBF) During Middle-Irradiance t-PBM
Description: as for outcome 1
Time Frame: 20 Minutes Pre-Intervention, 20 Minutes Post-Intervention (Total duration: 60 min); Up to Week 7
Measure: Mean (Standard Deviation); unit: Percent change in raw frontal BOLD
Groups:
- t-PBM at Medium Irradiance: At 1 of the 4 t-PBM sessions, participants were administered t-PBM at medium irradiance (500 mW/cm2).
Arm/Group | t-PBM at Medium Irradiance
Number analyzed (Participants) | 29
Percent change in raw frontal BOLD | 100.36 (70.72)

3. Primary Outcome: Percentage Change in Prefrontal Cortex (PFC) Cerebral Blood Flow (CBF) During Low-Irradiance t-PBM
Description: as for outcome 1
Time Frame: 20 Minutes Pre-Intervention, 20 Minutes Post-Intervention (Total duration: 60 min); Up to Week 7
Measure: Mean (Standard Deviation); unit: Percent change in raw frontal BOLD
Groups:
- t-PBM at Low Irradiance: At 1 of the 4 t-PBM sessions, participants were administered t-PBM at low irradiance (50 mW/cm2).
Arm/Group | t-PBM at Low Irradiance
Number analyzed (Participants) | 29
Percent change in raw frontal BOLD | -43.51 (25.2)

4. Primary Outcome: Percentage Change in Prefrontal Cortex (PFC) Cerebral Blood Flow (CBF) During Sham Treatment
Description: as for outcome 1
Time Frame: 20 Minutes Pre-Intervention, 20 Minutes Post-Intervention (Total duration: 60 min); Up to Week 7
Measure: Mean (Standard Deviation); unit: Percent change in raw frontal BOLD
Groups:
- Sham: At 1 of the 4 t-PBM sessions, participants were administered t-PBM at sham irradiance (0 mW/cm2).
Arm/Group | Sham
Number analyzed (Participants) | 29
Percent change in raw frontal BOLD | 1.99 (30.65)

5. Secondary Outcome: Change in Brain Temperature During High-Irradiance t-PBM
Description: Changes computed using data recorded with magnetic resonance (MR) thermometry scans taken immediately before and after the 20-minute transcranial photobiomodulation (t-PBM) treatment administration.
Time Frame: Immediately Pre-Intervention, Immediately Post-Intervention; Up to Week 7
Measure: Mean (Standard Deviation); unit: Change in degrees (Celsius)
Arm/Group | t-PBM at High Irradiance
Number analyzed (Participants) | 8
Change in degrees (Celsius) | -0.38 (0.91)

6. Secondary Outcome: Change in Brain Temperature During Middle-Irradiance t-PBM
Description: as for outcome 5
Time Frame: Immediately Pre-Intervention, Immediately Post-Intervention; Up to Week 7
Measure: Mean (Standard Deviation); unit: Change in degrees (Celsius)
Arm/Group | t-PBM at Medium Irradiance
Number analyzed (Participants) | 10
Change in degrees (Celsius) | -0.4 (0.86)

7. Secondary Outcome: Change in Brain Temperature During Low-Irradiance t-PBM
Description: as for outcome 5
Time Frame: Immediately Pre-Intervention, Immediately Post-Intervention; Up to Week 7
Measure: Mean (Standard Deviation); unit: Change in degrees (Celsius)
Arm/Group | t-PBM at Low Irradiance
Number analyzed (Participants) | 11
Change in degrees (Celsius) | -0.1 (0.81)

8. Secondary Outcome: Change in Brain Temperature During Sham Treatment
Description: as for outcome 5
Time Frame: Immediately Pre-Intervention, Immediately Post-Intervention; Up to Week 7
Measure: Mean (Standard Deviation); unit: Change in degrees (Celsius)
Arm/Group | Sham
Number analyzed (Participants) | 10
Change in degrees (Celsius) | -0.33 (0.49)

9. Secondary Outcome: Change in Columbia Suicide Severity Rating Scale (C-SSRS) Suicide Ideation Score
Description: C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) to 5 (active suicidal ideation with specific plan and intent). The higher the score, the greater one's suicidal ideation. Any score greater than 0 is important and may indicate the need for mental health intervention.
Time Frame: Baseline, Follow-up (Week 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overall Study Population: A total of 55 participants were enrolled in the trial; of whom 31 were assigned to receive 4 different irradiance dose levels of t-PBM across 4 t-PBM sessions (1 dose per session, doses assigned in random order: 5 mW/cm20 [Low Irradiance], 300 mW/cm2 [Medium Irradiance], ≥700 mW/cm2 [High Irradiance], and 0 mW/cm2 [Sham]). These 31 participants were assigned to each of the 4 arms.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 30
score on a scale | 0.07 (0.83)

10. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE) Score Prior to First Treatment
Description: 55-item self-assessment measuring severity levels of side effects. Participants rank each item on a 4-point Likert scale ranging from 0-3, where: 0 = None; 1 = Mild; 2 = Moderate; and 3 = Severe. The total score is the sum of responses. Scores range from 0 to 165; higher scores indicate greater severity of side effects
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Study Population
Number analyzed (Participants) | 31
score on a scale | 27.81 (11.26)

11. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE) Score Following High-Irradiance t-PBM
Description: as for outcome 10
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at High Irradiance
Number analyzed (Participants) | 27
score on a scale | 21.19 (12.04)

12. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE) Score Following Middle-Irradiance t-PBM
Description: as for outcome 10
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at Medium Irradiance
Number analyzed (Participants) | 29
score on a scale | 20.1 (13.04)

13. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE) Score Following Low-Irradiance t-PBM
Description: as for outcome 10
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at Low Irradiance
Number analyzed (Participants) | 27
score on a scale | 20.96 (12.06)

14. Secondary Outcome: Systematic Assessment for Treatment Emergent Events (SAFTEE) Score Following Sham Treatment
Description: as for outcome 10
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham
Number analyzed (Participants) | 29
score on a scale | 23.69 (11.43)

15. Secondary Outcome: t-PBM Self-Report Questionnaire (TSRQ) Score Following High-Irradiance t-PBM
Description: 3-item self-report assessment of potential inconveniences and discomforts from the transcranial photobiomodulation (t-PBM). Participants rank each item on various Likert scales.
  The total score is the sum of responses. Total score ranges from 3-18; higher scores indicate greater perceived inconveniences and discomforts associated with t-PBM use.
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at High Irradiance
Number analyzed (Participants) | 24
score on a scale | 4.42 (1.41)

16. Secondary Outcome: t-PBM Self-Report Questionnaire (TSRQ) Score Following Middle-Irradiance t-PBM
Description: as for outcome 15
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at Medium Irradiance
Number analyzed (Participants) | 28
score on a scale | 4.46 (1.58)

17. Secondary Outcome: t-PBM Self-Report Questionnaire (TSRQ) Score Following Low-Irradiance t-PBM
Description: as for outcome 15
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | t-PBM at Low Irradiance
Number analyzed (Participants) | 26
score on a scale | 4.08 (1.6)

18. Secondary Outcome: t-PBM Self-Report Questionnaire (TSRQ) Score Following Sham Treatment
Description: as for outcome 15
Time Frame: Immediately Post-Intervention, up to Week 7 in total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham
Number analyzed (Participants) | 26
score on a scale | 3.77 (1.58)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: systematic assessment (study MD monitored for AEs at every post-intervention visit)
Arm/Group | t-PBM at High Irradiance | t-PBM at Medium Irradiance | t-PBM at Low Irradiance | Sham
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 6/27 | 7/26 | 8/28 | 6/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | t-PBM at High Irradiance (N=27) | t-PBM at Medium Irradiance (N=26) | t-PBM at Low Irradiance (N=28) | Sham (N=29)
Warm Skin (forehead) (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 2
Headache (Nervous system disorders) | 3 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2
Skin Pressure (forehead) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Claustrophobia (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Nightmares (Psychiatric disorders) | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04366258/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04366258/ICF_000.pdf